CLINICAL TRIAL: NCT06052774
Title: The Effect of Non-Surgical Periodontal Therapy on Interleukin-34 in Stage I and II Periodontitis (A Controlled Clinical Trial With Biochemical Analysis)
Brief Title: Interleukin-34 in Stage I and II Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nada Zidan, teaching assistant in periodontology department- Ain shams University, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-Rec IR 092303
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cytokine Storm
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: Nonsurgical periodontal debridement was performed on patients using an ultrasonic scaler and universal curettes (2R - 2L and 4R- 4L). Oral Hygiene measures were instructed following treatment and follow-up after 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage I grade B periodontitis patients (Active Comparator): Nonsurgical periodontal debridement was performed on patients using an ultrasonic scaler and universal curettes (2R - 2L and 4R- 4L). Oral Hygiene measures were instructed following treatment and maintenance visits were given to them.
  Interventions: Procedure: Non-Surgical periodontal therapy
- Stage II grade B periodontitis patients (Active Comparator): Nonsurgical periodontal debridement was performed on patients using an ultrasonic scaler and universal curettes (2R - 2L and 4R- 4L). Oral Hygiene measures were instructed following treatment and maintenance visits were given to them.
  Interventions: Procedure: Non-Surgical periodontal therapy
- Periodontally healthy individuals (No Intervention): No intervention

INTERVENTIONS:
Procedure: Non-Surgical periodontal therapy — Supra and Subgingival debridement for all patients except periodontally healthy individuals
  Arms: Stage I grade B periodontitis patients; Stage II grade B periodontitis patients

SUMMARY:
Interleukin 34 (IL-34) is the second active component of (colony-stimulating factor receptor) CSF-1R. With regards to periodontal disease, It is debatable whether IL-34 is a pro-inflammatory cytokine (as seen in rheumatic arthritis and Sjogren syndrome) or an anti-inflammatory cytokine( as seen in Alzheimer's disease) so further studies could be conducted to better understand whether IL-34 is a proinflammatory or anti-inflammatory cytokine in the pathogenesis of periodontal diseases and to evaluate the change of its levels in Gingival crevicular fluid (GCF) in patients with periodontal disease after non-surgical periodontal therapy (NSPT).

DETAILED DESCRIPTION:
Periodontal disease is a multifactorial infection induced by a complex of bacterial species that interact with host tissues and cause destruction of the periodontal structures, including the supporting tissues of the teeth, alveolar bone, and periodontal ligament.

The bacterial biofilm formation initiates gingival inflammation; however, periodontitis initiation and progression depend on dysbiotic ecological changes in the microbiome in response to nutrients from gingival inflammatory and tissue breakdown products that enrich some species and anti-bacterial mechanisms that attempt to contain the microbial challenge within the gingival sulcus area once the inflammation has initiated.

Current evidence supports multifactorial disease influences, such as smoking, diabetes mellitus, obesity, metabolic syndrome, osteoporosis, low dietary calcium and vitamin D and other immunoinflammatory responses that make the dysbiotic microbiome changes more likely for some patients than others and likely influence the severity of disease for such individuals.

During periodontitis, the pathogen triggers the white blood cells of the innate immune system to release proinflammatory mediators such as cytokines that play a vital role in the progression of the inflammation process of periodontitis. In addition, these pathogens can activate the acquired immune system contributing to the release of more cytokines and chemokines that cause permanent bone damage and irreversible periodontal attachment loss.

Cytokines are defined as soluble small proteins (~5-20 kDa) that bind to specific receptors on certain cells, stimulate some internal cellular changes, and cause multiple genetic and chemical regulations.

There are two different types of inflammatory cytokines: proinflammatory cytokines that are involved in inflammatory reactions including interleukin-1 beta (IL-1β), interleukin-6 (IL-6), interleukin-12 (IL-12), tumor necrosis factor-alpha (TNF-α), and anti-inflammatory cytokines that regulate or control the pro-inflammatory cytokine response including interleukin-4 (IL-4), interleukin-1 receptor antagonist (IL-1RA) and interleukin-10 (IL-10).

NSPT aimed at the mechanical removal of bacterial plaque from the tooth surface is considered the "gold standard." This procedure decreases the number of Gram-negative bacteria in favor of Gram-positive bacteria as well as reduces the overall number of microorganisms in periodontal pockets and decreases the amount of proinflammatory cytokines.

Recent methods in oral and periodontal disease diagnostic research are identifying periodontal risk which is quantified by objective measures like biomarkers which are diagnostic tools to measure periodontal disease at the molecular, cellular, tissue, and clinical levels. The biological media for detecting periodontal disease biomarkers include GCF, saliva, serum, subgingival plaque, and tissue biopsies.

The major attraction of GCF as a diagnostic marker is the site-specific nature of the sample which may offer the basis for patient-specific diagnostic tests for periodontal disease. Moreover, the simplicity of its use along with a level of reliability and low cost favors its use over other modalities.

The discovery of new biomarkers will aid in the development of new therapeutic approaches via host modulatory drugs for periodontal disease treatment leading to more individualized, targeted treatments for oral health.

In 2008, Lin identified a secreted protein known as IL-34 with a high functional selectivity represented by stimulating monocyte survival in a CSF-1R-dependent manner. Many studies provided insight into IL-34 biology, but many questions remain unanswered, specifically in terms of its function.

High expression of IL-34 correlates with disease severity in autoimmune diseases (Sjögren's syndrome, SLE, and RA), and inflammatory diseases (liver fibrosis, kidney disease, and inflammatory bowel disease). In contrast, IL-34 plays a protective role in some diseases, such as atopic dermatitis, Alzheimer's disease, breast cancer, and head and neck cancer.

In periodontal disease, some studies such as Guruprasad & Pradeep in 2018 and Bozkurt Doğan in 2021 suggested that IL-34 is a proinflammatory cytokine in the pathogenesis of periodontal disease while others such as Martinez in 2017 and Lira-Junior in 2021 concluded that IL-34 play a protective role in periodontal disease.

Therefore, Further studies must be carried out to confirm these findings and to better understand the possible role of IL-34 in the pathogenesis of periodontal diseases and to evaluate its levels in GCF in patients with periodontal disease after NSPT

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage I and II grade B Periodontitis in addition to periodontally healthy individuals.
* Both genders aged from 20-50 years
* Minimum 20 natural teeth excluding third molars.
* Good compliance with the plaque control instructions following initial therapy.
* Availability for follow-up and maintenance program.

Exclusion Criteria:

* Smokers.
* Pregnant and lactating females.
* Systemic diseases that could affect the outcome of the therapy (According to the Cornell Medical Index-Health Questionnaire).
* Patients taking antibiotics, anti-inflammatory drugs, and immunosuppressive therapy during the preceding 6 months before the start of the trial and during the study.
* Patients who have undergone any periodontal therapy in the last 6 months.
* Vulnerable groups of patients' e.g. (handicapped patients).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
To measure the IL - 34 levels in GCF before &after NSPT of stage I and II grade B periodontitis patients in comparison to periodontally healthy individuals | 3 months
  To measure the IL - 34 levels in ng/L before &after NSPT of stage I and II grade B periodontitis patients in comparison to periodontally healthy individuals

SECONDARY OUTCOMES:
To evaluate Plaque index before & after NSPT in Stage I and II grade B periodontitis patients | 3 months
  To evaluate Plaque index (0 score indicated zero plaque to 3 score that indicated highest plaque index score) before & after NSPT in Stage I and II grade B periodontitis patients
To evaluate Gingival index before & after NSPT in Stage I and II grade B periodontitis patients | 3 months
  To evaluate Gingival index (0 score indicated no bleeding to 3 score that indicated excessive bleeding ) before & after NSPT in Stage I and II grade B periodontitis
To evaluate probing depth before & after NSPT in Stage I and II grade B periodontitis | 3 months
  To evaluate probing depth (in mm) before & after NSPT in Stage I and II grade B periodontitis
To evaluate Clinical attachment Level before & after NSPT in Stage I and II grade B periodontitis | 3 months
  To evaluate Clinical attachment Level (in mm) before & after NSPT in Stage I and II grade B periodontitis

CONTACTS AND LOCATIONS:
Overall Officials: hala A. Abuel Ela, Professor, Study Director — Professor of Oral Medicine, Periodontology, Oral Diagnosis, Faculty of Dentistry, ASU; Doaa Adel-Khattab, Asso.Prof., Study Chair — Associate Prof. of oral medicine, Periodontology and Oral diagnosis Faculty of dentistry ASU
Locations (1):
- Faculty of Dentistry-Ain Shams University, Cairo, Egypt

REFERENCES:
- See also: Serum cytokine levels in periodontitis patients in relation to the bacterial load — http://pubmed.ncbi.nlm.nih.gov/21138356/
- See also: Gingival Crevicular Fluid (GCF): A Diagnostic Tool for the Detection of Periodontal Health and Diseases — http://pubmed.ncbi.nlm.nih.gov/33668185/
- See also: Emerging roles of Interleukin-34 together with receptor activator of nuclear factor-kB ligand and — http://pubmed.ncbi.nlm.nih.gov/34034144/
- See also: Tooth loss in complying and non-complying periodontitis patients with different periodontal risk levels during supportive periodontal care — http://pubmed.ncbi.nlm.nih.gov/33760975/
- See also: Diagnostic potential and future directions of biomarkers in gingival crevicular fluid and saliva of periodontal diseases: Review of the current evidence — http://pubmed.ncbi.nlm.nih.gov/29288920/
- See also: Effect of nonsurgical periodontal therapy on interleukin-34 levels in periodontal health and disease — http://pubmed.ncbi.nlm.nih.gov/29900909/
- See also: Periodontitis: A Multifaceted Disease of Tooth-Supporting Tissues — http://pubmed.ncbi.nlm.nih.gov/31370168/
- See also: Discovery of a cytokine and its receptor by functional screening of the extracellular proteome — http://pubmed.ncbi.nlm.nih.gov/18467591/
- See also: Levels of myeloid-related proteins in saliva for screening and monitoring of periodontal disease — http://pubmed.ncbi.nlm.nih.gov/34409624/
- See also: Salivary Colony Stimulating Factor-1 and Interleukin-34 in Periodontal Disease — http://pubmed.ncbi.nlm.nih.gov/28474967/
- See also: Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions — http://pubmed.ncbi.nlm.nih.gov/29926490/
- See also: Staging and grading of periodontitis: Framework and proposal of a new classification and case definition — http://pubmed.ncbi.nlm.nih.gov/29926952/
- See also: Cytokines, inflammation, and pain — http://pubmed.ncbi.nlm.nih.gov/17426506/